CLINICAL TRIAL: NCT02929940
Title: Multi-center Study of the Liver Disease in European Patients With alpha1-antitrypsin Deficiency
Brief Title: Liver Disease in Patients With alpha1-antitrypsin Deficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: Alpha1-Liver
Record Dates: First submitted 2016-10-06; First posted 2016-10-11 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: alpha1-antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood specimen for serologic and genetic analyses
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- PiZZ: Observational
  Interventions: Other: No intervention
- PiMZ: Observational
  Interventions: Other: No intervention
- Other AATD variants: Observational
  Interventions: Other: No intervention
- PiMM (Control): Observational
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No Intervention, observational

SUMMARY:
Alpha1-antitrypsin deficiency (AATD) is the third most common genetic disorder leading to death worldwide. Apart from lung disease, AATD also leads to liver involvement in up to 50% of patients. Hence, liver involvement is the second most common cause of morbidity and mortality in AATD patients. But the natural history of disease in adults is not well understood and specific therapies are still in the phase of preclinical studies. Despite these facts and the therapeutic and preventative potential, the AATD-related liver disease is still largely being neglected by both the patients and the healthcare professionals.

To improve the hepatologic care of patients with AATD, the investigators initiated a prospective multi-center study in Europe that systematically evaluates the liver function in these patients and their relatives. The investigators cooperate with both patient organizations as well as with lung centers specialized on AATD-related lung disease.

DETAILED DESCRIPTION:
Alpha1-antitrypsin deficiency (AAT deficiency) is a frequently overlooked metabolic disorder. Apart from lung disease, AAT deficiency also leads to liver disease. This can affect people of all ages and all ethnic groups. Although involvement of the liver is the second most common cause of decreased quality of life and life expectancy in Alpha1 patients, no preventative care plan, like that one implemented to avoid lung involvement, has yet been drawn up.

Chronic liver involvement therefore often remains undetected until a very late stage in diagnosed cases of AAT deficiency. This is compounded by the fact that the patients affected generally have only unspecific symptoms if any at all. Moreover, routine diagnostic measurements (e.g. liver function tests) often reveal no abnormalities. In the case of a late diagnosis, the diverse complications of liver disease can no longer be effectively prevented.

Liver involvement in AAT deficiency can lead to liver cirrhosis or liver cancer. Liver cirrhosis is the life-threatening consequence of many liver disorders and carries a poor prognosis. Besides AAT deficiency, many other - potentially treatable - conditions, such as viral hepatitis, excessive alcohol consumption and diabetes, can cause liver damage. Liver cirrhosis itself leads to many, often life-threatening secondary disorders such as heavy bleeding or liver cancer. It is therefore crucial that liver disorders such as AAT deficiency are diagnosed at an early stage, so as to prevent complications and to treat concomitant risk factors.

The investigators collaborate with various patient support groups and other hospitals specialising in AAT deficiency-associated lung disease. Together with their collaborators, the investigators hope to improve the care of affected patients and help to bring about therapeutic advances.

The aim of this study is to clarify how liver function is modified in patients with AAT deficiency. For this, among other things, the investigators use:

(i) modern ultrasound-based scanners for non-invasive measurement of the degree of liver scarring.

(ii) Specialized liver parameters in blood samples, which also provide information on any existing liver disorders (iii) Questionnaire.

Study participants receive a full, cost-free analysis of their individual liver involvement and are given appropriate recommendations for disease prevention. The examinations provide a relief to many and to everybody,the investigators are able to offer an individual liver damage prevention plan.

All adult patients (of every genotype) as well as any family members interested will be studied and advised. Besides the specialist clinic in Aachen (Germany), free examinations throughout and even outside of Germany will be offered.

ELIGIBILITY:
Inclusion Criteria:

* All patients with known AATD (every genotype)
* Relatives of patients with known AATD

Exclusion Criteria:

* Children
* Pregnant women
* Patients who cannot give informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with alpha1-antitrypsin deficiency (AATD) and their relatives.
  AATD is the third most common genetic disorder leading to death worldwide. Apart from lung disease, AATD also leads to liver involvement in up to 50% of patients. Hence, liver involvement is the second most common cause of morbidity and mortality in AATD patients. The natural history of disease is not well understood and specific therapies are lacking. Accordingly, the AATD-related liver disease is still largely being neglected by both the patients and the healthcare professionals.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-04; Primary Completion 2020-04 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Liver fibrosis, Hepatic decompensation, Liver cancer, Death or Liver transplantation | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Strnad, MD, Principal Investigator — RWTH Aachen University
Locations (1):
- RWTH Aachen University, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spivak I, Guldiken N, Usachov V, Schaap F, Damink SWMO, Bouchecareilh M, Lehmann A, Fu L, Mo FR, Ensari GK, Hufnagel F, Fromme M, Preisinger C, Strnad P. Alpha-1 Antitrypsin Inclusions Sequester GRP78 in a Bile Acid-Inducible Manner. Liver Int. 2025 Jan;45(1):e16207. doi: 10.1111/liv.16207. PMID 39665869
- [Derived] Hamesch K, Mandorfer M, Pereira VM, Moeller LS, Pons M, Dolman GE, Reichert MC, Schneider CV, Woditsch V, Voss J, Lindhauer C, Fromme M, Spivak I, Guldiken N, Zhou B, Arslanow A, Schaefer B, Zoller H, Aigner E, Reiberger T, Wetzel M, Siegmund B, Simoes C, Gaspar R, Maia L, Costa D, Bento-Miranda M, van Helden J, Yagmur E, Bzdok D, Stolk J, Gleiber W, Knipel V, Windisch W, Mahadeva R, Bals R, Koczulla R, Barrecheguren M, Miravitlles M, Janciauskiene S, Stickel F, Lammert F, Liberal R, Genesca J, Griffiths WJ, Trauner M, Krag A, Trautwein C, Strnad P; European Alpha1-Liver Study Group. Liver Fibrosis and Metabolic Alterations in Adults With alpha-1-antitrypsin Deficiency Caused by the Pi*ZZ Mutation. Gastroenterology. 2019 Sep;157(3):705-719.e18. doi: 10.1053/j.gastro.2019.05.013. Epub 2019 May 20. PMID 31121167
- See also: Alpha1-Liver Website (German) — http://www.alpha1-leber.de
- See also: Alpha1-Liver Website (English) — http://www.alpha1-liver.eu